CLINICAL TRIAL: NCT06568497
Title: Sensory, Satiating and Glycaemic Characteristics of Cheese and Non-dairy Alternative Products to Cheese
Brief Title: Dairy and Vegan Cheese: Effect on Satiety and Blood Glucose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023-147
Record Dates: First submitted 2024-08-01; First posted 2024-08-23 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Blood Glucose; Satiety Response
MeSH Terms: interventions — Food

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dairy (Experimental): A food containing dairy cheese
  Interventions: Other: Food
- Non-Dairy (Experimental): A food containing vegan alternative to cheese
  Interventions: Other: Food
- Conrtol (Experimental): A control treatment in the form of food
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Food

SUMMARY:
The project will consist of two studies. One study will explore the satiating properties of dairy cheese and its dairy-free substitute when consumed ad libidum, and another study will investigate their effects on postprandial glycemia. Both studies will involve healthy young adults. The secondary outcomes of these studies will be food sensory characteristics, diet-induced thermogenesis, subjective feeling of fatigue and energy, gastrointestinal comfort level, and food intake. The proposed project results will help to better understand the health properties of the cheese and its dairy-free substitute.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy adults

Exclusion Criteria:

* Breakfast skipper
* Smoker (including e-cigarettes) / cannabis consumer
* Be underweight, overweight or obese
* Have chronic diseases, including diabetes
* Taking certain medication
* Have lactose intolerance, food allergies or gastrointestinal disorders (e.g., irritable bowel syndrome, or others).

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-08-04 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | 0-120 minutes
  The concentrations of blood glucose
Insulin | 0-120 minutes
  The concentrations of insulin
Satiety | 0-120 minutes
  The components of average subjective appetite including desire to eat, hunger, fullness, and a prospective food consumption measured with 100mm visual analogue scales.
Food intake | 0 minutes, 120 minutes
  Energy intake with an ad libitum meal at 120 minutes

SECONDARY OUTCOMES:
Energy and Fatigue | 0-120 minutes
  Subjective perception of feeling energetic and fatigue
Gastrointestinal comfort | 0-120 minutes
  The subjective feeling of wellness and gastrointestinal discomfort parameters including the feeling of nausea, stomach cramps, flatulency, diarrhea and a subjective feeling of wellness, each measured with 100mm visual analogue scales.
Diet-induced thermogenesis | 0-120 minutes
  Indirect calorimetry
Sensory characteristics | 0 minutes, 120 minutes
  The perception of pleasantness of the treatments (0 minutes) and a test meal (at 120 minutes) will be measured with 9-point hedonic and 100mm visual analogue scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No